CLINICAL TRIAL: NCT01117584
Title: Phase 2b, Double-Blind, Randomized, Multicenter, Parallel Group, Placebo-Controlled, Dose-Finding Study to Evaluate the Efficacy, Safety and Tolerability of a 12-Week Treatment With ASP1941 in Combination With Metformin in Patients With Type 2Diabetes Mellitus Who Have Inadequate Glycemic Control on Metformin Alone
Brief Title: A Study to Evaluate the Effect of ASP1941 in Combination With Metformin in Adult Patients With Type 2 Diabetes Mellitus
Acronym: BALANCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1941-CL-0005; 2009-013881-25 (EudraCT Number)
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes; ASP1941; diabetes; metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — ipragliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- ASP1941 lowest dose (Experimental): oral tablet
  Interventions: Drug: ipragliflozin; Drug: Metformin
- ASP1941 low dose (Experimental): oral tablet
  Interventions: Drug: ipragliflozin; Drug: Metformin
- ASP1941 high dose (Experimental): oral tablet
  Interventions: Drug: ipragliflozin; Drug: Metformin
- ASP1941 highest dose (Experimental): oral tablet
  Interventions: Drug: ipragliflozin; Drug: Metformin
- Placebo (Placebo Comparator): oral tablet
  Interventions: Drug: Placebo; Drug: Metformin

INTERVENTIONS:
Drug: ipragliflozin — oral tablet
  Other Names: ASP1941
  Arms: ASP1941 high dose; ASP1941 highest dose; ASP1941 low dose; ASP1941 lowest dose
Drug: Placebo — oral tablet
  Arms: Placebo
Drug: Metformin — oral tablet

SUMMARY:
Evaluate the efficacy, safety and tolerability of a 12-week treatment of 4 doses of ASP1941 compared to placebo in combination with metformin in adult patients with Type 2 Diabetes Mellitus who have inadequate glycemic control on metformin alone.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been diagnosed with Diabetes Mellitus type 2 (T2DM) for at least 6 months
* Subject has inadequate glycemic control indicated by an HbA1c level between 7.0% and 9.5% at start of the run-in period at Visit 1 AND does not meet any of the FPG discontinuation criteria
* Subject has been on a stable dose of at least 1500 mg/day metformin monotherapy for at least 6 weeks prior to Visit 1
* Subject is on a stable diet and exercise program (for at least 6 weeks prior to Visit 1) and is willing to remain on this program for the duration of the study
* Subject has a body mass index (BMI) 20 - 45 kg/m2 at Visit 1
* Female subject of childbearing potential has a negative serum pregnancy test (human chorionic gonadotropin [hCG]) at Visit 1 and agrees to use an acceptable form of contraception throughout the duration of the study OR is at least 1 year post-menopausal (defined as amenorrhea for at least 1 year) or surgically sterile. Male study subjects should be advised to use a male condom in addition to having their partner use another acceptable method during the study and for 3 months after the last dose

Exclusion Criteria:

* Subject has any known complication of T2DM indicating a late disease state that in the investigator's opinion should preclude the subject from participation
* Subject has type 1 diabetes mellitus
* Subject is in need of insulin therapy or has received insulin within 3 months prior to Visit 1, with the exception of acute use of <7 days
* Subject has a serum creatinine higher than upper limit of normal range at Visit 1
* Subject has an alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) higher than 3 times upper limit of normal range or has a total bilirubin more than 2 times upper limit of normal at Visit 1
* Subject has a urinary microalbumin/creatinine ratio above or equal to 300 mg/g at Visit 1
* Subject has a symptomatic urinary tract infection (UTI) or symptomatic genital infection at Visit 1 or during the placebo run-in period, including just prior to randomization at Visit 2
* Subject has persistent, uncontrolled severe hypertension as indicated by a systolic blood pressure >180 mmHg or a diastolic blood pressure of >110 mmHg taken in a sitting position after 5 minutes of rest on at least 2 measurements (within 30 minutes of each other) at Visit 1
* Subject has a significant cardiovascular disease, such as myocardial infarction or a vascular intervention (e.g. angioplasty or stent) within 3 months prior to Visit 1, or history of heart failure (New York Heart Association [NYHA] Class III IV)
* Subject is known to have hepatitis or be a carrier of hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody (enzyme linked immunosorbent assay [ELISA] plus confirmatory test), or is known positive for human immunodeficiency virus (HIV) HIV-1 and/or HIV 2
* Subject is currently receiving an excluded medication (loop-diuretics or systemic corticosteroids) or has received any other oral anti-diabetic drug except for metformin within 3 months prior to Visit 1
* Subject has history of lactic acidosis
* Subject has a history of drug or alcohol abuse/dependency within 12 months prior to Visit 1 as defined in the Diagnostic and Statistical Manual-IV (DSM-IV)
* Subject has had a malignancy in the last 5 years, except for adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Female subject who is pregnant, lactating or pre-menopausal with positive serum pregnancy test (hCG) at Visit 1 or has an intention of becoming pregnant
* Subject has an unstable medical or psychiatric illness
* Subject has known or suspected hypersensitivity to ASP1941 or any components of the formulations used
* Subject has previously received ASP1941
* Subject is concurrently participating in another drug study or has received an investigational drug within 30 days (or the limit set by national law, whichever is longer) prior to Visit 1
* Subject has any concurrent illness which, in the opinion of the investigator, may interfere with treatment or evaluation of safety or completion of this study
* In the investigator's judgment, the subject is unable to adhere to the treatment regimen, protocol procedures or study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2010-04-06 (Actual); Primary Completion 2011-04-01 (Actual); Study Completion 2011-04-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at Week 12 | Baseline, 12 weeks

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose (FPG) at Week 12 | Baseline, 12 weeks
Achievement of target goal (HbA1c <7.0%) at Week 12 | 12 weeks
Achievement of target goal (HbA1c <6.5%) at Week 12 | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ude Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (34):
- United States (5):
  - Los Angeles, California
  - Coral Gables, Florida
  - Hialeah, Florida
  - Kissimmee, Florida
  - Las Vegas, Nevada
- Hungary (7):
  - Baja
  - Balatonfüred
  - Budapest
  - Gyöngyös
  - Makó
  - Nyíregyháza
  - Zalaegerszeg
- Italy (3):
  - Ancona
  - Milan
  - Siena
- Poland (8):
  - Chrzanów
  - Katowice
  - Krakow
  - Kutno
  - Lodz
  - Lublin
  - Warsaw
  - Wroclaw
- Romania (7):
  - Brasov
  - Bucharest
  - Constanța
  - Craiova
  - Lasi
  - Ploieşti
  - Sibiu
- United Kingdom (4):
  - Birmingham
  - Cambridgeshire
  - Manchester
  - Reading

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Kashiwagi A, Shestakova MV, Ito Y, Noguchi M, Wilpshaar W, Yoshida S, Wilding JPH. Safety of Ipragliflozin in Patients with Type 2 Diabetes Mellitus: Pooled Analysis of Phase II/III/IV Clinical Trials. Diabetes Ther. 2019 Dec;10(6):2201-2217. doi: 10.1007/s13300-019-00699-8. Epub 2019 Oct 12. PMID 31606880
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=2